CLINICAL TRIAL: NCT04438460
Title: Pediatric Immune Response to Multi-Organ Dysfunction
Acronym: PedIMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_0068; 2020-A00343-36 (Other: ID-RCB)
Record Dates: First submitted 2020-05-28; First posted 2020-06-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multiple Organ Dysfunction Syndrome
Keywords: Multiple organ dysfunction; Immunosuppression; mHLA-DR; Pediatrics; Secondary infection
MeSH Terms: conditions — Multiple Organ Failure; Coinfection | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): 150 children aged 1 month to 12 years with multi-visceral failure syndrome within 48 hours of hospitalization in pediatric resuscitation will be included in this study
  Interventions: Biological: Blood test
- Control group (Other): 60 children aged 1 month to 12 years hospitalized for simple elective surgery will be included in this study
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — For patient group, blood tests will be performed at day 1-2, day 3-5 and day 60.
  For control group, blood test will be performed the day of elective surgery.

SUMMARY:
Multiple organ dysfunction (MOD) is defined by the association of at least two failures of vital organs, with various etiologies (septic shock, polytrauma, acute respiratory distress syndrome, etc.). Associated mortality remains high in children (between 20 and 50%).

In septic shock, one of the main causes of MOD, induced immunosuppression can occur, with immune alterations affecting all cells of immunity. This induced immunosuppression is associated with an additional risk of secondary acquired infections and death in adults. Among all the cells and all the markers studied, the expression of Human Leukocyte Antigen - DR isotype (HLA-DR) on the surface of the monocyte (mHLA-DR, expressed in number of sites per cell) appeared as one of the best biomarkers of this induced immunosuppression. Decreased expression of monocyte Human Leukocyte Antigen - DR isotype (mHLA-DR) in adults is linked to an increased risk of developing secondary infection and death.

These results were confirmed by team in the context of pediatric septic shock, with an attack of innate immunity in the foreground. Persistent lowering of mHLA-DR for more than 3 days after onset of shock was associated with the occurrence of secondary acquired infections: 50% of children had mHLA-DR of less than 8000 sites / cells on D3, of which 60 % developed secondary infection within 30 days. No child with mHLA-DR greater than 8000 sites / cells had secondary infection.

Such immune alterations appear to be non-specific for septic shock, as they have also been described after multiple trauma or severe respiratory infections.

The hypothesize is that multi-systemic aggression leading to multi-visceral failure syndrome could also lead to significant immunosuppression, regardless of the etiology of this MOD.

At present, the proportion of persistent immunosuppression induced by MOD, all etiologies combined, is poorly documented in pediatrics. Estimating this proportion in a large pediatric cohort, while exploring as fully as possible the associated immune alterations and acquired secondary infections, would improve the pathophysiological understanding and pediatric specificities of this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

Patient Group:

* 1 month < Age < 12 years
* Multiple organ dysfunction within 48 hours following intensive care unit admission
* Beneficiary of a social security scheme.
* Consent signed by at least one parent / holder of parental authority

Control Group:

* 1 month < Age < 12 years
* Hospitalized for simple elective surgery
* Beneficiary of a social security scheme.
* Consent signed by at least one parent / holder of parental authority

Exclusion Criteria:

Patient Group:

* Weight < 5 kg
* Known immunosuppression
* Prolonged corticotherapy
* Chronic inflammatory disease
* Malignant pathology with ongoing treatment
* Hepatic cirrhosis
* Polymerase Chain Reaction (PCR) Severe acute respiratory syndrome coronavirus (SARS-CoV-2) positive or patient with Pediatric Inflammatory Multisystem Syndrome (PIMS)
* Pediatric inflammatory multisystem syndrome (PIMS)

Control Group:

* Weight < 5 kg
* Known immunosuppression
* Prolonged corticotherapy
* Chronic inflammatory disease
* Malignant pathology with ongoing treatment
* Ongoing infection
* Organ failure
* Hepatic cirrhosis
* PCR SARS-CoV-2 positive or patient with Pediatric Inflammatory Multisystem Syndrome (PIMS)
* Pediatric inflammatory multisystem syndrome (PIMS)

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Secondary acquired infection (SAI) | Day 60
  This criterion will be related to the duration of follow-up and expressed as an incidence of SAI occurrence.This incidence will be calculated in the two groups "Presence of immunosuppression" and "Absence of immunosuppression", defined from the value of mHLA-DR at D3-D5: "Presence of immunosuppression" if mHLA-DR < 8000 sites/cells and "Absence of immunosuppression" if mHLA-DR ≥ 8000 sites/cells. The diagnosis of secondary acquired infection will be made by an independent committee.

SECONDARY OUTCOMES:
blood counts : Characterization of alterations in the myeloid lineage | Day 1
  Blood cell counts will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
mHLA-DR expression : Characterization of alterations in the myeloid lineage | Day 1
  mHLA-DR expressed as a number of site / cell will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months
transcriptome : Characterization of alterations in the myeloid lineage | Day 1
  Gene expression through messenger ribonucleic acid (mRNA) analysis will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
plasma cytokines : Characterization of alterations in the myeloid lineage | Day 1
  Cytokine levels will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
blood counts : Characterization of alterations in the myeloid lineage | Day 3
  Blood cell counts will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months
mHLA-DR expression : Characterization of alterations in the myeloid lineage | Day 3
  mHLA-DR expressed as a number of site / cell will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
transcriptome : Characterization of alterations in the myeloid lineage | Day 3
  Gene expression through messenger ribonucleic acid (mRNA) analysis will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
plasma cytokines : Characterization of alterations in the myeloid lineage | Day 3
  Cytokine levels will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
blood counts : Characterization of alterations in the myeloid lineage | Day 60
  Blood cell counts will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
mHLA-DR expression : Characterization of alterations in the myeloid lineage | Day 60
  mHLA-DR expressed as a number of site / cell will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
transcriptome : Characterization of alterations in the myeloid lineage | Day 60
  Gene expression through messenger ribonucleic acid (mRNA) analysis will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
plasma cytokines : Characterization of alterations in the myeloid lineage | Day 60
  Cytokine levels will be compared between the groups "secondary acquired infections" and "no secondary acquired infection" occurring within 2 months.
mHLA-DR measurement | Day 60
  Evaluation of the immunological recovery at month 2 with regard to the initial state and in comparison with the controls.
Myeloid Derived Suppressor Cells (MDSC) measurement | Day 1
  Characterization of MDSC will be measured and compared between patient and control
Intra-cellular production of tumor necrosis factor alpha (TNFα) by the monocyte | Day 1
  Evaluate the feasibility of a new test : measure of the intra-cellular production of TNF α by the monocyte. It will be compared between patient and control.
MDSC measurement | Day 3
  Characterization of MDSC will be measured
Intra-cellular production of TNFα by the monocyte | Day 3
  Evaluate the feasibility of a new test : measure of the intra-cellular production of TNF α by the monocyte.
Monocytic and dendritic subpopulations measurement | Day 1
  Characterization of monocytic and dendritic subpopulations will be realized and compared between patient and control.
Gamma-delta T lymphocytes measurement | Day 1
  Characterization of gamma-delta T lymphocytes will be realized and compared between patient and control.
Monocytic and dendritic subpopulations measurement | Day 3
  Characterization of monocytic and dendritic subpopulations will be realized
Gamma-delta T lymphocytes measurement | Day 3
  Characterization of gamma-delta T lymphocytes will be realized
Monocytic and dendritic subpopulations measurement | Day 60
  Characterization of monocytic and dendritic subpopulations will be realized
Gamma-delta T lymphocytes measurement | Day 60
  Characterization of gamma-delta T lymphocytes will be realized

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant, Bron
  - Hopital Mère Enfant, Nantes